CLINICAL TRIAL: NCT01871727
Title: A Clinical Study to Demonstrate Safety and Efficacy of E7777 in Persistent or Recurrent Cutaneous T-Cell Lymphoma
Brief Title: A Trial of E7777 in Persistent and Recurrent Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Dr. Reddy's Laboratories Limited (Industry); Citius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7777-G000-302
Record Dates: First submitted 2013-03-28; First posted 2013-06-07 (Estimated); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2022-11

CONDITIONS: Persistent or Recurrent Cutaneous T-Cell Lymphoma
Keywords: Persistent or Recurrent Cutaneous T-Cell Lymphoma; E7777
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E7777 (Experimental)
  Interventions: Drug: E7777 9 mcg/kg

INTERVENTIONS:
Drug: E7777 9 mcg/kg — administered by intravenous (i.v.) infusion over 60 minutes (+/-10 minutes) on 5 consecutive days during every cycle of 21 days

SUMMARY:
The purpose of this trial is to assess the efficacy of E7777 in participants with recurrent or persistent Cutaneous T-Cell Lymphoma (CTCL) in Stage I - III participants as assessed by objective response rate (ORR). A lead-in dose-finding part was used to determine dose level 9 microgram per kilogram (mcg/kg) E7777 that is being used to test efficacy and safety.

DETAILED DESCRIPTION:
This is a multicenter, open-label study of E7777 in participants with recurrent or persistent CTCL. The study consists of an initial Lead-in part (to select recommended dose of E7777 for Main part), followed by the Main part (to test efficacy). Participants will move through three phases while on study: Pretreatment Phase, Treatment Phase, and Extension Phase and a Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in the study:

1. Age greater than or equal to 18 years.
2. Histopathologic diagnosis of CTCL (mycosis fungoides [MF] or Sezary Syndrome [SS]), confirmed by skin biopsy, or lymph node, or blood assessment, of current disease.
3. CD25 assay-positive tumor, defined as detectable CD25 on greater than or equal to 20% of total lymphoid infiltrate in biopsied lesions by immunohistochemistry.
4. CTCL disease stage at study entry as follows, according to ISCL/EORTC (Olsen 2011).

   * Lead-In Part: Stage IA - IV, except participants with CNS involvement.
   * Main Study: Stage I - III
5. History of prior therapies for CTCL: must have had prior therapy, any number of prior therapies allowed.

   Topical treatments (except topical chemotherapy) and steroids are not considered as prior therapies.
6. A minimum washout period of 4 weeks after previous CTCL therapy is recommended before the first dose of E7777.

   Participants must have recovered from any adverse effects from any previous CTCL therapy to Common Terminology Criteria for Adverse Events (CTCAE) Grade <2 before starting study drug. A shorter washout may be allowed if participant is experiencing progressive disease despite ongoing treatment.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 in the Lead-In Part and performance status of 0 or 1 in the Main Study.
8. Life expectancy greater than or equal to 3 months in the Lead-In Part and greater than or equal to 12 months in the Main Study.
9. Adequate bone marrow reserves as evidenced by:

   * platelets greater than or equal to 100,000/mm^3 (100 x 10^9/L)
   * clinically stable hemoglobin greater than or equal to 9 gram per deciliter (g/dL) (90 g/L) and hematocrit greater than or equal to 27% without transfusion support
10. Normal hepatic function as evidenced by:

    * bilirubin <= 1.5* upper limit if normal (ULN) and alkaline phosphatase <=3.0*ULN
    * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3.0*ULN
    * albumin >= 3.0 g/dL (30 g/L)
11. Adequate renal function as evidenced by serum creatinine less than or equal to 1.8 mg/dL (158 umol/L) or calculated creatinine clearance greater than or equal to 50 mL/min (per the Cockcroft-Gault formula) with less than 2+ protein or 24- hour urine creatinine clearance greater than or equal to 50 mL/minute with 24- hour urine protein less than 1gram.
12. Provide written informed consent prior to any study-specific screening procedures.
13. Females may not be lactating or pregnant at Screening or Baseline
14. All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically
15. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partner must meet the criteria above

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from the study:

1. Prior denileukin diftitox therapy
2. Use of topical steroids within 14 days of Day 1 of initial therapy is not allowed.Topical steroids or systemic low dose steroids of less than or equal to 10 milligram per day (mg/day) prednisone are allowed in participants with erythroderma who have been on corticosteroids for a prolonged period of time and where discontinuation may lead to rebound flare in disease. The concomitant steroid medication is allowed as long as the type of steroid, route of administration, and steroid dose remain the same as what the participant had been receiving for a prolonged period of time.
3. Active malignancy (except for CTCL, definitively treated basal or squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix) within the past 24 months.
4. Serious intercurrent illness
5. Significant cardiac disease requiring ongoing treatment, including congestive heart failure (CHF), severe coronary artery disease (CAD), cardiomyopathy, uncontrolled cardiac arrhythmia, unstable angina pectoris, or myocardial infarction (MI)
6. Significant pulmonary symptoms or disease
7. History of uncontrolled seizure disorder or active central nervous system disease
8. Major surgery within 2 weeks of study enrollment
9. Significant or uncontrolled infections requiring systemic anti-infective therapy
10. Known human immunodeficiency virus (HIV) infection; known active hepatitis B or hepatitis C infection
11. Females who are pregnant (positive urine test) or breastfeeding
12. Any history of a medical condition or a concomitant medical condition that, in the opinion of the investigator, would compromise the participant's ability to safely complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (18):
  - University of Alabama at Birmingham, Dermatology at Whitaker Clinic, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Medical Center National Medical Center, Duarte, California
  - UC Irvine Health-Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford University Cancer Center, Stanford, California
  - Yale University Cancer Center, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of PittsburghMedical Center Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of TX MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Epworth Healthcare Freemasons, East Melbourne, Victoria
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico

REFERENCES:
- [Derived] Foss FM, Kim YH, Prince HM, Akilov OE, Querfeld C, Seminario-Vidal L, Fisher DC, Kuzel TM, Yannakou CK, Geskin LJ, Feldman T, Sokol L, Allen PB, Dang NH, Cabanillas F, Wong HK, Ooi CE, Xing D, Sauter N, Singh P, Czuczman M, Duvic M. Efficacy and Safety of Denileukin Diftitox-Cxdl, an Improved Purity Formulation of Denileukin Diftitox, in Patients With Relapsed or Refractory Cutaneous T-Cell Lymphoma. J Clin Oncol. 2025 Apr;43(10):1198-1209. doi: 10.1200/JCO-24-01549. Epub 2024 Dec 19. PMID 39700456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in the United States and Australia from 30 May 2013 to 14 December 2021.
Pre-assignment Details: 36 participants were screened in Lead-In Part, out of which 21 were enrolled and treated.143 participants were screened in Main Study Part, out of which 91 were enrolled and 90 were treated. As per planned analysis, data was collectively reported for total 98 participants (Full analysis set/Safety analysis set) from Main Study Part and Lead-In Part who received study drug at 9 micrograms per kilograms (mcg/kg) dose. 8 participants were from Lead-In Part and 90 were from Main Study Part.
Groups:
- Lead-In Part: E7777 6 mcg/kg: Participants were treated with E7777 6 mcg/kg by intravenous (IV) infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part.
- Lead-In Part: E7777 9 mcg/kg: Participants were treated with E7777 9 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part.
- Lead-In Part: E7777 12 mcg/kg: Participants were treated with E7777 12 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part.
- Lead-In Part: E7777 15 mcg/kg: Participants were treated with E7777 15 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-In Part.
- Main Study Part: E7777 9 mcg/kg: Participants were treated with E7777 9 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Main study part.
Period: Lead-In Part (1 Year 2 Months)
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg | Main Study Part: E7777 9 mcg/kg
Started | 2 | 8 | 9 | 2 | 0
Primary Efficacy Analysis Set | 0 | 5 (The primary efficacy analysis set was defined as participants who had Stage I to III Cutaneous T-Cell Lymphoma (CTCL) at baseline and received E7777 at 9 mcg/kg; this set included 64 participants from the Main Study and 5 participants from the Lead-In part- this set had total 69 participants.) | 0 | 0 | 0
Completed | 1 | 4 | 5 | 2 | 0
Not Completed | 1 | 4 | 4 | 0 | 0
Not completed — Disease Progression | 1 | 4 | 4 | 0 | 0
Period: Main Study Part (2 Years 4 Months)
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg | Main Study Part: E7777 9 mcg/kg
Started | 0 | 0 | 0 | 0 | 91
Primary Efficacy Analysis Set | 0 | 0 | 0 | 0 | 64 (The primary efficacy analysis set was defined as participants who had Stage I to III Cutaneous T-Cell Lymphoma (CTCL) at baseline and received E7777 at 9 mcg/kg; this set included 64 participants from the Main Study and 5 participants from the Lead-In part- this set had total 69 participants.)
Completed | 0 | 0 | 0 | 0 | 46
Not Completed | 0 | 0 | 0 | 0 | 45
Not completed — Other | 0 | 0 | 0 | 0 | 2
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 9
Not completed — Disease progression | 0 | 0 | 0 | 0 | 20
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Not treated | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Lead-In Part: Safety Analysis Set (SAS) included all participants who received study drug. Main Study Part: SAS included all participants (both Main Study and Lead-In) who received study drug at 9 mcg/kg. As per planned analysis baseline data was collected and reported for 98 participants who received 9 mcg/kg dose in lead-in and main study part.
Groups:
- Lead-In Part: E7777 6 mcg/kg: Participants were treated with E7777 6 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part.
- Lead-In Part and Main Study Part: E7777 9 mcg/kg: Participants were treated with E7777 9 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part and in Main study part and were presented together here, as planned.
- Total: Total of all reporting groups
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg | Lead-In Part and Main Study Part: E7777 9 mcg/kg | Total
Number analyzed (Participants) | 2 | 9 | 2 | 98 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (22.63) | 58.4 (15.88) | 69.0 (2.83) | 62.9 (11.91) | 62.5 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 37 | 45
  Male | 0 | 5 | 0 | 61 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 14 | 15
  Not Hispanic or Latino | 2 | 8 | 2 | 81 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 16 | 20
  White | 1 | 7 | 1 | 73 | 82
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Lead-In Part: Number of Participants With Dose-limiting Toxicities (DLTs) as Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03)
Description: DLTs as per NCI CTCAE v4.03 were defined as 1) serious infusion reaction (CTCAE) Grade 4 adverse event of "Infusion related reaction," or recurrent CTCAE Grade 3 despite administration of systemic steroid premedication after initial occurrence. Infusion reactions were defined as symptoms (example, fatigue, nausea, vomiting, arthralgia, myalgia, pyrexia, chills, rigors) occurring within 24 hours of E7777 infusion. 2) Capillary leak syndrome (CLS) CTCAE Grade 4 or Grade 3 (with exceptions). A CLS event was defined as the noted occurrence of at least 2 of the following: hypotension, edema, or serum albumin less than (<) 3.0 gram per decilitre (g/dL). 3) Clinical visual impairment. 4) Any CTCAE Grade greater than or equal to (>=) 4 adverse event (AE) that may represent an infusion reaction. 5) Any other Grade 3 or greater toxicity assessed as related to E7777 treatment and which in the opinion of a safety consultancy investigator panel, was a dose-limiting toxicity.
Time Frame: Cycle 1 (cycle length was 21 days)
Population: Lead-in analysis set included all participants enrolled in lead-in part.
Measure: Count of Participants; unit: Participants
Groups:
- Lead-In Part: E7777 9 mcg/kg: Participants were treated with E7777 9 mcg/kg by IV infusion over 60 minute on 5 consecutive days during every 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-In Part.
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 8 | 9 | 2
Participants | 0 | 0 | 0 | 2

2. Primary Outcome: Lead-In Part: Maximum Tolerated Dose (MTD) of E7777
Description: The MTD was defined as the safe dose level established in Lead-In Part. MTD was determined by summarizing the number and percentage of participants with DLTs for the first cycle, by study dosing schedule, initial dosing level and overall for the Lead-In Part.
Time Frame: Cycle 1 (cycle length was 21 days)
Population: Dose-finding analysis set included all participants in the Lead-in part who completed Cycle 1 treatment and were evaluated for DLT, and those who discontinued during Cycle 1 due to DLT.
Measure: Number; unit: mcg/kg
Groups:
- Lead-In Part: E7777: Participants were treated with E7777 6, 9, 12 and 15 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-In part.
Arm/Group | Lead-In Part: E7777
Number analyzed (Participants) | 21
mcg/kg | 12.0

3. Primary Outcome: Main Study Part: Objective Response Rate (ORR) by Independent Review Committee (IRC) Based on Olsen 2011 Criteria
Description: ORR was defined as the percentage of participants whose best overall response (BOR) was complete response (CR) or partial response (PR) based on independent review committee on 2 assessments at least 3 weeks apart. The tumor response was based on global response score (GRS) Olsen 2011 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites.
Time Frame: From the date of administration of the first dose of the study drug until disease progression (Up to 3 years 6 months)
Population: Primary efficacy analysis set included all participants with Stages I to III CTCL (both Main Study and Lead-In part) who received study drug at the 9 mcg/kg dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Main Study Part: E7777 9 mcg/kg: Participants with stages I to III CTCL were treated with E7777 9 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part and in Main study part and were presented together here, as planned.
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 69
percentage of participants | 36.2 [25.0 to 48.7]

4. Secondary Outcome: Lead-In Part: Duration of Response (DOR) Per Investigator Assessment
Description: DOR per investigator assessment was defined as the time from date when criteria for response (CR or PR) was first met until the date of the first documentation of disease progression (PD) or date of death from any cause. The tumor assessment was based on GRS Olsen 2011 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites. PD was defined as any new lesion or unequivocally increase of previously involved sites from nadir.
Time Frame: From the date of first documentation of CR or PR until date of the first documentation of PD or death due to any cause (Up to 1 year 2 months)
Population: Lead-in analysis set included all participants enrolled in the Lead-in part. Here, 'overall number of participants analyzed' were those who had CR or PR in lead in part.
Measure: Median (Full Range); unit: days
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 1 | 4 | 3 | 0
days | 43.0 [43 to 43] | 106.0 [71 to 134] | 113.0 [92 to 351] |

5. Secondary Outcome: Main Study Part: Duration of Response (DOR) Per Independent Review Committee
Description: DOR per independent review committee was defined as the time from the date when criteria for response (CR or PR) was first met until the date of the first documentation of PD or date of death from any cause. The tumor assessment was based on GRS Olsen 2011 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites. PD was defined as any new lesion or unequivocally increase of previously involved sites from nadir.
Time Frame: From the date of first documentation of CR or PR until date of the first documentation of PD or death due to any cause (Up to 3 years 6 months)
Population: Primary efficacy analysis set included all participants with Stages I to III CTCL (both Main Study and Lead-In part) who received study drug at the 9 mcg/kg dose. Here, 'overall number of participants analyzed' were those who had CR or PR in Lead-in part and in Main study part.
Measure: Median (Full Range); unit: months
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 25
months | 6.47 [3.0 to 23.5]

6. Secondary Outcome: Lead-In Part: Time to Response (TTR) Per Investigator Assessment
Description: Time to response per investigator assessment was defined as the time from date of first dose to the date of the first documented CR or PR. The tumor assessment was based on GRS Olsen 2011 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites.
Time Frame: From the date of administration of the first dose of the study drug until date of the first documentation of PR or CR (Up to 1 year 2 months)
Population: Lead-in analysis set included all participants enrolled in the Lead-in part. Here, 'overall number of participants analyzed' were those who had CR or PR in lead-in part of the study.
Measure: Median (Full Range); unit: days
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 1 | 4 | 3 | 0
days | 106.0 [106.0 to 106.0] | 53.5 [22 to 85] | 64.0 [57 to 106] |

7. Secondary Outcome: Main Study Part: Time to Response (TTR) Per Independent Review Committee
Description: Time to response per independent review committee was defined as the time from date of first dose to the date of the first documented CR or PR. The tumor assessment was based on GRS Olsen 2011 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites.
Time Frame: From the date of administration of the first dose of the study drug until date of the first documentation of PR or CR (Up to 3 years 6 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 25
months | 1.41 [0.7 to 5.6]

8. Secondary Outcome: Lead-In Part and Main Study Part: ORR Per Investigator Assessment
Description: ORR per investigator assessment was defined as the percentage of participants whose BOR was CR or PR. The tumor response was based on GRS Olsen 2011 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites.
Time Frame: From the date of administration of the first dose of the study drug until disease progression (Up to 3 years 6 months)
Population: Lead-in analysis set included all participants enrolled in the lead-in part and Investigator efficacy analysis set included all Stage I to III participants (both Main Study [n=66] and Lead-In [n=5]) who received study drug at 9 mcg/kg dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 2 | 8 | 9 | 2 | 71
percentage of participants | 50.0 [1.3 to 98.7] | 50.0 [15.7 to 84.3] | 33.3 [7.5 to 70.1] | 0 [0 to 84.2] | 42.3 [30.6 to 54.6]

9. Secondary Outcome: Main Study Part: ORR Per IRC Based on Prince 2010 Criteria
Description: ORR was defined as the percentage of participants whose BOR was CR, clinical complete response (CCR) or PR per IRC. The tumor response was based on Prince 2010 criteria. CR was defined as disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites. CCR was defined as tumor residue not visible on esophagogram, computed tomography (CT), endoscopy, positron emission tomography (PET)-CT.
Time Frame: From the date of administration of the first dose of the study drug until disease progression (Up to 3 years 6 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 69
percentage of participants | 36.2 [25.0 to 48.7]

10. Secondary Outcome: Lead-In Part and Main Study Part: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was defined as an adverse event that had an onset date, or a worsening in severity on or after the first dose of study drug up to the end of the study. SAE was any untoward medical occurrence that at any dose: resulted in death; life threatening required inpatient hospitalization; resulted in persistent, significant disability; was congenital anomaly/birth defect or medically important due to other reasons than mentioned criteria. Number of participants with TEAEs and SAEs were reported.
Time Frame: From the first dose of study drug up to 30 days after the last dose (Up to 3 years and 7 months)
Population: Lead-In Part: SAS included all participants who received study drug. Main Study Part: SAS included all participants (both Main Study and Lead-In) who received study drug at 9 mcg/kg.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg | Lead-In Part and Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 2 | 9 | 2 | 98
Participants
  TEAEs | 2 | 9 | 2 | 97
  SAEs | 0 | 4 | 2 | 36

11. Secondary Outcome: Lead-In Part: Maximum Serum Concentration (Cmax) of E7777
Description: Participants were not available for analysis in 15 mcg/kg (Cycles 3 and 5), 6 mcg/kg (Cycle 5), 9 mcg/kg (Cycles 3 and 5), 12 mcg/kg (Cycle 3), hence no Pharmacokinetic (PK) data was collected and analyzed for these doses and cycles.
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 minutes post-dose (Cycle length was 21 days)
Population: Lead-in PK analysis set included all participants who received at least one dose of study drug and from whom at least one valid E7777 PK parameter was obtained. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure for given timepoints.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Lead-In Part: E7777 9 mcg/kg: Participants were treated with E7777 9 mcg/kg by IV infusion over 60 minutes on 5 consecutive days during every 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-In Part.
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 7 | 8 | 2
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 135 (26.2) | 118 (70.8) | 183 (65.3) | 383 (133)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 59.5 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 105 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |

12. Secondary Outcome: Main Study Part: Maximum Serum Concentration (Cmax) of E7777
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 minutes post-dose (Cycle length was 21 days)
Population: Main study part PK analysis set included all participants from whom at least one quantifiable concentration of E7777 was observed at 9 mcg/kg dose (both Main Study and Lead-In). Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 20
ng/mL
  Cycle 1 Day 1 | 114 (62.5)
  Cycle 3 Day 1: number analyzed (Participants) | 16
  Cycle 3 Day 1 | 37.5 (19.4)
  Cycle 5 Day 1: number analyzed (Participants) | 12
  Cycle 5 Day 1 | 45.5 (46.8)

13. Secondary Outcome: Lead-In Part: Area Under the Curve From Time 0 to Time t (AUC[0-t]) of E7777
Description: Participants were not available for analysis in 15 mcg/kg (Cycles 3 and 5), 6 mcg/kg (Cycle 5), 9 mcg/kg (Cycles 3 and 5), 12 mcg/kg (Cycle 3), hence no PK data was collected and analyzed for these doses and cycles. Here, min*ng/mL means minute*nanogram per milliliter.
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 hours Post-dose (Cycle length was 21 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 7 | 8 | 2
min*ng/mL
  Cycle 1 Day 1 | 18500 (6080) | 18200 (13100) | 23600 (12900) | 39800 (4170)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 4670 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 6730 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |

14. Secondary Outcome: Main Study Part: Area Under the Curve From Time 0 to Time t (AUC[0-t]) of E7777
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: Main study part PK analysis set included all participants from whom at least one quantifiable concentration of E7777 was observed at 9 mcg/kg dose (both Main Study and Lead-In). Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 20
min*ng/mL
  Cycle 1 Day 1 | 16300 (12600)
  Cycle 3 Day 1: number analyzed (Participants) | 16
  Cycle 3 Day 1 | 2170 (974)
  Cycle 5 Day 1: number analyzed (Participants) | 12
  Cycle 5 Day 1 | 2660 (2570)

15. Secondary Outcome: Lead-In Part: Area Under the Curve From Time 0 to Time Infinity (AUC[0-inf]) of E7777
Description: Participants were not available for analysis in 15 mcg/kg (Cycles 3 and 5), 6 mcg/kg (Cycle 5), 9 mcg/kg (Cycles 3 and 5), 12 mcg/kg (Cycle 3), hence no PK data was collected and analyzed for these doses and cycles.
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 4 | 5 | 1
min*ng/mL
  Cycle 1 Day 1 | 20600 (7850) | 27000 (16500) | 30000 (12900) | 43500 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis.
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 4960 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 6900 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |

16. Secondary Outcome: Main Study Part: Area Under the Curve From Time 0 to Time Infinity (AUC[0-inf]) of E7777
Description: Participants were not available for analysis at Cycle 3 Day 1, hence no PK data was collected and analyzed for this timepoint.
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 10
min*ng/mL
  Cycle 1 Day 1 | 23700 (12700)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 4630 (NA) — Standard deviation could not be estimated for Cycle 5 Day 1 as insufficient number of participants were available for analysis.

17. Secondary Outcome: Lead-In Part: Terminal Elimination Half-life (t1/2) of E7777
Description: as for outcome 15
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: minutes
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 4 | 5 | 2
minutes
  Cycle 1 Day 1 | 92.0 [74.5 to 109] | 116 [55.9 to 138] | 100 [47.9 to 120] | 100 [71.5 to 129]
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 39.6 [39.6 to 39.6] |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 20.5 [20.5 to 20.5] |

18. Secondary Outcome: Main Study Part: Terminal Elimination Half-life (t1/2) of E7777
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 14
Measure: Median (Full Range); unit: minutes
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 12
minutes
  Cycle 1 Day 1 | 109 [58.9 to 168]
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1 | 90.8 [90.8 to 90.8]
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 51.7 [51.7 to 51.7]

19. Secondary Outcome: Lead-In Part: Time to Reach Maximum (Peak) Concentration After Drug Administration (Tmax)
Description: as for outcome 15
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: minute
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 7 | 8 | 2
minute
  Cycle 1 Day 1 | 75 [60 to 90] | 60 [30 to 180] | 61.5 [49.2 to 90] | 60 [60 to 60]
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 60 [60 to 60] |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 60 [60 to 60] |

20. Secondary Outcome: Main Study Part: Time to Reach Maximum (Peak) Concentration After Drug Administration (Tmax)
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 14
Measure: Median (Full Range); unit: minutes
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 20
minutes
  Cycle 1 Day 1 | 60 [28 to 180]
  Cycle 3 Day 1: number analyzed (Participants) | 16
  Cycle 3 Day 1 | 60 [30 to 74]
  Cycle 5 Day 1: number analyzed (Participants) | 12
  Cycle 5 Day 1 | 60 [30 to 64]

21. Secondary Outcome: Lead-In Part: Total Body Clearance (CL) of E7777
Description: Participants were not available for analysis in 15 mcg/kg (Cycles 3 and 5), 6 mcg/kg (Cycle 5), 9 mcg/kg (Cycles 3 and 5), 12 mcg/kg (Cycle 3), hence no PK data was collected and analyzed for these doses and cycles. Here, mL/min/kg means milliliter per minute per kilogram.
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 4 | 5 | 1
mL/min/kg
  Cycle 1 Day 1 | 0.316 (0.12) | 0.492 (0.38) | 0.551 (0.48) | 0.359 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis.
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 1.21 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 1.80 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |

22. Secondary Outcome: Main Study Part: Total Body Clearance (CL) of E7777
Description: as for outcome 16
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: Main study part PK analysis set included all participants from whom at least one quantifiable concentration of E7777 was observed at 9 mcg/kg dose (both Main Study and Lead-In). Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure for given time points.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 10
mL/min/kg
  Cycle 1 Day 1 | 44.6 (32.6)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 133 (NA) — Standard deviation could not be estimated for Cycle 5 Day 1 as insufficient number of participants were available for analysis.

23. Secondary Outcome: Lead-In Part: Volume of Distribution at Steady State (Vdss) of E7777
Description: as for outcome 15
Time Frame: Cycles 1, 3, 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 4 | 5 | 1
milliliter per kilogram (mL/kg)
  Cycle 1 Day 1 | 39.8 (4.81) | 60.3 (19.50) | 61 (21.80) | 37 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis.
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 3 Day 1 | 69.1 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 5 Day 1 |  |  | 53.3 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis. |

24. Secondary Outcome: Main Study Part: Volume of Distribution at Steady State (Vdss) of E7777
Description: as for outcome 16
Time Frame: Cycles 1, 3 and 5 Day 1: Pre-dose up to 300 hours post-dose (Cycle length was 21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 20
milliliter (mL)
  Cycle 1 Day 1 | 5430 (2210)
  Cycle 3 Day 1: number analyzed (Participants) | 0
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 10700 (NA) — Standard deviation could not be estimated for Cycle 5 Day 1 as insufficient number of participants were available for analysis.

25. Secondary Outcome: Lead-In Part: Percentage of Participants Testing Positive for Anti-E7777 and Anti-interleukin (IL)-2 Antibodies
Description: Immunogenicity was assessed by determining the anti-E7777 and anti-IL-2 antibodies in serum using validated methods. Percentage of participants testing positive for Anti-E7777 and Anti-IL-2 antibodies were reported.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 5 Day 1
Population: Lead-in PK Analysis Set included all participants who received at least one dose of study drug and from whom at least one valid E7777 PK parameter was obtained.
Measure: Number; unit: percentage of participants
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 9 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg
Number analyzed (Participants) | 2 | 8 | 9 | 2
percentage of participants
  Cycle 1 Day 1 (Anti-E7777 Antibodies) | 50.0 | 100.0 | 88.9 | 100.0
  Cycle 2 Day 1 (Anti-E7777 Antibodies) | 100.0 | 100.0 | 83.3 | 0
  Cycle 3 Day 1 (Anti-E7777 Antibodies) | 100.0 | 100.0 | 100.0 | 0
  Cycle 5 Day 1 (Anti-E7777 Antibodies) | 100.0 | 100.0 | 100.0 | 0
  Cycle 1 Day 1 (Anti-IL-2 Antibodies) | 0 | 37.5 | 33.3 | 0
  Cycle 2 Day 1 (Anti-IL-2 Antibodies) | 0 | 87.5 | 83.3 | 0
  Cycle 3 Day 1 (Anti-IL-2 Antibodies) | 100.0 | 100.0 | 100.0 | 0
  Cycle 5 Day 1 (Anti-IL-2 Antibodies) | 100.0 | 83.3 | 100.0 | 0

26. Secondary Outcome: Main Study Part: Percentage of Participants Testing Positive for Anti-E7777 and Anti-IL-2 Antibodies
Description: as for outcome 25
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1
Population: Main Study Part PK Analysis Set included all participants from whom at least one quantifiable concentration of E7777 was observed at 9 mcg/kg dose (both Main Study and Lead-In).
Measure: Number; unit: percentage of participants
Groups:
- Main Study Part: E7777 9 mcg/kg: Participants were treated with E7777 9 mcg/kg by IV infusion over 60 minutes on 5 consecutive days in 21-day cycles for up to 8 cycles or disease progression or unacceptable toxicity in Lead-in part and in Main study part and were presented together here, as planned.
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 94
percentage of participants
  Cycle 1 Day 1 (Anti-E7777 Antibodies) | 85.7
  Cycle 2 Day 1 (Anti-E7777 Antibodies) | 91.7
  Cycle 3 Day 1 (Anti-E7777 Antibodies) | 95.7
  Cycle 1 Day 1 (Anti-IL-2 Antibodies) | 5.5
  Cycle 2 Day 1 (Anti-IL-2 Antibodies) | 52.3
  Cycle 3 Day 1 (Anti-IL-2 Antibodies) | 88.6

27. Secondary Outcome: Main Study Part: Number of Participants With Objective Skin Response
Description: Modified severity weighted assessment tool (mSWAT) was used to measure skin disease severity based on the percentage of body surface area (BSA) with patches, plaques, or tumors. Total scores were calculated by multiplying the BSA percentage for each category of lesion (patch, plaque, or tumor) by a weighting factor and adding the three sub-scores which ranged from 0 (unaffected) to 400 (severely affected). Lower scores indicated a lower degree of skin disease severity. CR corresponded to 100% clearance of skin lesions present at baseline (mSWAT score of 0). PR corresponded to 50-99% clearance of skin disease present at baseline (at least 50% reduction in mSWAT score), without new tumors.
Time Frame: Up to 30 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 69
Participants | 25

28. Secondary Outcome: Main Study Part: Duration of Skin Response
Description: The duration of skin response based on the mSWAT score was defined as time from the date when criteria for skin response (CR or PR) was first met until the date of documented PD or death due to any cause for those participants with a confirmed PR or CR. mSWAT was used to measure skin disease severity based on the percentage of BSA with patches, plaques, or tumors. Total scores were calculated by multiplying the BSA percentage for each category of lesion (patch, plaque, or tumor) by a weighting factor and adding the three sub-scores which ranged from 0 (unaffected) to 400 (severely affected). Lower scores indicated a lower degree of skin disease severity. CR corresponded to 100% clearance of skin lesions present at baseline (mSWAT score of 0). PR corresponded to 50-99% clearance of skin disease present at baseline (at least 50% reduction in mSWAT score), without new tumors.
Time Frame: Up to 30 months
Population: Primary efficacy analysis set included all participants with Stages I to III CTCL (both Main Study and Lead-In part) who received study drug at the 9 mcg/kg dose. Here 'overall number of participants analyzed' were those who had a skin response.
Measure: Median (Full Range); unit: months
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 25
months | 6.47 [3.0 to 23.5]

29. Secondary Outcome: Main Study Part: Time to Skin Response
Description: The time to skin response based on the mSWAT score was defined as time from the date of first dose to the date when criteria for skin response (CR or PR) were first met. mSWAT was used to measure skin disease severity based on the percentage of BSA with patches, plaques, or tumors. Total scores were calculated by multiplying the BSA percentage for each category of lesion (patch, plaque, or tumor) by a weighting factor and adding the three sub-scores which ranged from 0 (unaffected) to 400 (severely affected). Lower scores indicated a lower degree of skin disease severity. CR corresponded to 100% clearance of skin lesions present at baseline (mSWAT score of 0). PR corresponded to 50-99% clearance of skin disease present at baseline (at least 50% reduction in mSWAT score), without new tumors.
Time Frame: Up to 30 months
Population: as for outcome 28
Measure: Median (Full Range); unit: months
Arm/Group | Main Study Part: E7777 9 mcg/kg
Number analyzed (Participants) | 25
months | 1.41 [0.7 to 5.6]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose (Up to 3 years and 7 months)
Description: Lead-In Part: SAS included all participants who received study drug. Main Study Part: SAS included all participants (both Main Study and Lead-In) who received study drug at 9 mcg/kg. As per planned analysis,all participants from lead-in part (9 mcg/kg) arm were reported together with the main study part participants (98=9 participants from 9 mcg/kg lead-in part and 90 participants from main study part) hence, data was reported for 98 participants as planned in main study part for this section.
Arm/Group | Lead-In Part: E7777 6 mcg/kg | Lead-In Part: E7777 12 mcg/kg | Lead-In Part: E7777 15 mcg/kg | Lead-In Part and Main Study Part: E7777 9 mcg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 3/9 | 0/2 | 13/98
Serious Adverse Events (participants affected / at risk) | 0/2 | 4/9 | 2/2 | 36/98
Other Adverse Events (participants affected / at risk) | 2/2 | 9/9 | 1/2 | 95/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-In Part: E7777 6 mcg/kg (N=2) | Lead-In Part: E7777 12 mcg/kg (N=9) | Lead-In Part: E7777 15 mcg/kg (N=2) | Lead-In Part and Main Study Part: E7777 9 mcg/kg (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 3
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 3
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 8
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 2 | 11
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-In Part: E7777 6 mcg/kg (N=2) | Lead-In Part: E7777 12 mcg/kg (N=9) | Lead-In Part: E7777 15 mcg/kg (N=2) | Lead-In Part and Main Study Part: E7777 9 mcg/kg (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 8
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 6
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 5
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 5
Dry eye (Eye disorders) | 1 | 0 | 0 | 6
Vision blurred (Eye disorders) | 0 | 0 | 0 | 8
Eye inflammation (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 6
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 0 | 15
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 19
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 0 | 38
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 12
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 26
Fatigue (General disorders) | 1 | 6 | 0 | 29
Generalised oedema (General disorders) | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 0 | 28
Pain (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 15
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Pustule (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 10
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 19
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0 | 27
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 26
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 7
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Respiratory rate decreased (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 14
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 6
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 10
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 9
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 18
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 14
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 5
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 16
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 7
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 6
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0 | 9
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT01871727/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT01871727/SAP_001.pdf